CLINICAL TRIAL: NCT00572390
Title: Oestrogen Withdrawal in Hypopituitary Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Jens Sandahl Christiansen, Århus universityhospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: oestrogen withdrawal; 1999/4644
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2007-12

CONDITIONS: Hypopituitarism
MeSH Terms: conditions — Hypopituitarism | interventions — Estrogens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): No oestrogen treatment
  Interventions: Drug: oestrogen
- 2 (Experimental): Oestrogen treatment
  Interventions: Drug: oestrogen

INTERVENTIONS:
Drug: oestrogen — Cyclic oestrogen substitution therapy

SUMMARY:
By exploring hormonal status in hypopituitary women during oestrogen treatment and without estrogen substitution the influence on sexhormones and organ function is estimated.

DETAILED DESCRIPTION:
38 hypopituitary women were examinined twice. During oestrogen treatment and after 1 month estrogen withdrawal. A control group of healthy women were examined once.Antropometric data and hormonal parameters were collected.

ELIGIBILITY:
Inclusion Criteria:

* Hypopituitarism

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2001-01; Study Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
androgens, IGF-I, body composition, liver enzymes, | 1 month

SECONDARY OUTCOMES:
Grehlin, adiponection, leptin | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jens J Christiansen, PhD, Principal Investigator — Århus Universityhospital
Locations (1):
- Århus Universityhospital, Aarhus, Denmark

REFERENCES:
- [Derived] Host C, Christiansen JJ, Christiansen JS, Jorgensen JO, Gravholt CH. Discontinuation of hormone replacement therapy in young GH-treated hypopituitary women increases liver enzymes. Growth Horm IGF Res. 2010 Feb;20(1):26-30. doi: 10.1016/j.ghir.2009.07.001. Epub 2009 Aug 5. PMID 19660970